CLINICAL TRIAL: NCT04904198
Title: A Care Management Intervention for Non-cardiac Chest Pain: Intervention Development and Feasibility Assessment
Brief Title: A Care Management Intervention for Non-cardiac Chest Pain
Acronym: NCCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Associate Chief of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P002331
Record Dates: First submitted 2021-05-18; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Chest Pain
Keywords: non-cardiac chest pain; atypical chest pain; collaborative care
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Care Management Intervention for Non-cardiac chest pain (Experimental): Multicomponent care management intervention.
  Interventions: Behavioral: Care Management Intervention for non-cardiac chest pain

INTERVENTIONS:
Behavioral: Care Management Intervention for non-cardiac chest pain — Multicomponent eight-week care management intervention involving a consultation visit with a cardiologist and nurse. Recommendations from the consultation visit are conveyed to the primary care physician. Following the visit, the participant has eight weekly phone calls with a nurse to provide support, introduce therapeutic principals, and assess symptoms. The study nurse is supervised by a psychiatrist.

SUMMARY:
The investigators developed and implemented an eight-week multicomponent care management intervention for non-cardiac chest pain. Team members including a cardiologist, nurse, and psychiatrist. Impressions and recommendations were shared with the patient's primary care physician. Measures of chest pain severity, frequency and impact and measures of psychological health and health-related quality of life were completed at baseline and intervention completion.

DETAILED DESCRIPTION:
The investigators developed and implemented an eight-week multicomponent care management intervention for non-cardiac chest pain. The care management team consisted of a nurse, cardiologist, and psychiatrist. Following a one-time consultation visit with the cardiologist and nurse, evaluation and treatment recommendations were conveyed to the participant's primary care physician. Then, the nurse completed eight weekly phone calls with the participant to provide support, introduce therapeutic principles, and assist with coordination of care, under the supervision of a psychiatrist. Intervention feasibility was assessed on several domains including adherence, recruitment, attrition, safety, and data collection. To examine preliminary efficacy, participants completed Likert scales of chest pain symptom severity, frequency and impact, and measures of psychological health (Patient Health Questionnaire-9, General Anxiety Disorder-7, Patient Health Questionnaire-15) and health-related quality of life (12-Item Short Form Survey) at baseline and intervention completion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-cardiac chest pain, defined as chest pain recurring at least once per week for two weeks with at least two of the following objective tests: (1) electrocardiogram without ischemic changes; (2) negative cardiac enzymes; (3) non-ischemic cardiac stress test.
* Primary care physician affiliated with the institution

Exclusion Criteria:

* History or subsequent diagnosis of cardiac disease
* Objectively diagnosed alternative medical etiology of chest pain (e.g., gastroesophageal disease)
* Resolution of chest pain prior to enrollment
* Cognitive impairment, assessed using a six-item screen
* Inability to communicate in English
* Lack of telephone access (precluding weekly phone call participation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of adherence | Week 8
  A priori, feasible adherence was defined as 100% completion of the consultation visit and a mean completion of at least half of the eight phone calls over the eight-week study period.

SECONDARY OUTCOMES:
Feasibility of recruitment | Baseline
  Collect data on the proportion of individuals interested in the study who meet eligibility criteria for participation
Feasibility of intervention attrition | Week 8
  A priori, an attrition rate of less than or equal to 15% was defined as indicating intervention feasibility
Feasibility of intervention safety | Week 8
  Any adverse psychological or physical symptoms were documented throughout the study intervention with appropriate follow-up to ensure safety
Feasibility of data collection at baseline | Baseline
  Assessment of whether participants would be able to complete all baseline study measures
Feasibility of data collection at follow-up | Week 8
  Assessment of whether participants would be able to complete all follow-up study measures
Change in chest pain symptom severity | Change from baseline at week 8
  Likert scale from 0 (no pain) to 10 (severe pain)
Change in chest pain symptom frequency | Change from baseline at week 8
  Likert scale from 0 (infrequent) to 10 (very frequent)
Change in chest pain symptom impact | Change from baseline at week 8
  Likert scale from 0 (no impact) to 10 (severe impact)
Change in depressive symptoms | Change from baseline at week 8
  Patient Health Questionnaire-9, score range of 0-27, higher numbers reflect more severe symptoms.
Change in anxiety symptoms | Change from baseline at week 8
  General Anxiety Disorder-7, score range of 0-21, higher numbers reflect more severe symptoms.
Change in somatic symptom disorder/somatization symptoms | Change from baseline at week 8
  Patient Health Questionnaire-15, score range of 0-30, higher numbers reflect more severe symptoms.
Change in health-related quality of life | Change from baseline at week 8
  12-Item Short Form Survey. Generates a physical health composite summary and a mental health composite summary. The mean score is set to 50 for each composite score. Scores > 50 indicate better physical or mental health-related quality of life than the mean, and scores < 50 indicate worse physical or mental health-related quality of life than the mean.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Jeff Huffman, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madva EN, Celano CM, Kim S, Bell M, Radfar A, Ibrahim NE, Dar T, Albanese A, Tawakol A, Huffman JC. A Care Management Intervention for Noncardiac Chest Pain: Treatment Development and Feasibility Assessment. Prim Care Companion CNS Disord. 2022 Apr 19;24(2):21m03045. doi: 10.4088/PCC.21m03045. PMID 35452569